CLINICAL TRIAL: NCT03198039
Title: Guided Meditation as an Adjunct to Enhance Postoperative Recovery: A Feasibility Study
Brief Title: Guided Meditation as an Adjunct to Enhance Postoperative Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2017P000239
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Feasibility of a Meditation Program Perioperatively
Keywords: Meditation; Cognitive Dysfunction; Postoperative Period; Cardiac Surgery
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Meditation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Meditation twice daily for at least two weeks prior to surgery and for four weeks after surgery
  Interventions: Behavioral: Meditation
- Group 2 (Experimental): Meditation twice daily for four weeks after surgery
  Interventions: Behavioral: Meditation
- Group 3 (No Intervention): Control group - will undergo surgery and subsequent hospital stay according to the current standard of care, which does not include meditation

INTERVENTIONS:
Behavioral: Meditation — Isha Kriya (IK) meditation approximately 12 minutes, twice a day
  Arms: Group 1; Group 2

SUMMARY:
The primary purpose of this trial is to test the feasibility of implementing a meditation program in the perioperative period.

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled study involving 30 adult patients undergoing cardiac surgery. Investigators will test the feasibility of implementing a meditation program in the perioperative period. Patients will be randomized to one of three groups: those who complete Isha Kriya (IK) meditation before and after surgery, those who complete postoperative IK meditation only, and those who receive the standard of care with no meditation intervention. In addition to testing feasibility, the investigators will explore whether a meditation program can affect recovery after surgery. Patients enrolled will be followed postoperatively for up to one month to assess their cognitive function, pain, and sleep. Blood will also be collected for analysis of biomarkers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Undergoing any of the following types of cardiac surgery: CABG with or without valve surgery (aortic and/or mitral); isolated valve surgery; isolated aortic surgery
3. Surgery scheduled for at least 14 days after enrollment

Exclusion Criteria:

1. Urgent and/or emergent surgery
2. Non-English speaking
3. Cognitive impairment as defined by total MoCA score < 10
4. Baseline DASS-21 depression score >10
5. Pre-existing history of psychiatric illness as documented in the medical record or divulged in history taking in pre-enrollment patient interview, such as anxiety, depression, or bipolar disorder
6. History of cerebrovascular accident or recent history (< 3 months) of seizures
7. History of dementia, Parkinson's disease, Alzheimer's disease, or other forms of cognitive decline
8. Current use of cognition enhancing drugs
9. Current management for chronic pain
10. Currently enrolled in another interventional study that could impact the primary outcome, as determined by the PI
11. Educational attainment below high school level or equivalent
12. Significant visual impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2017-11-28 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Adherence to implementing a meditation program in the perioperative period | Baseline through 1 month post surgery
  In this descriptive, feasibility study, evaluation of feasibility will include adherence to meditation intervention (total number of sessions completed).

SECONDARY OUTCOMES:
Cognitive function - MoCA | Baseline and hospital discharge (approximately 5 days)
  The Montreal Cognitive Assessment (MoCA) will be administered at baseline and hospital discharge. This is a validated test that measures cognitive impairment.
Pain scores | Postoperative Day 1 through hospital discharge (approximately 5 days)
  Postoperative pain will be assessed with a standard 11-point scale. Pain scores will be obtained by asking the subject.
Total Opioid Consumption | Intraoperatively through 48 hours postoperatively
  The total opioid dosage received in the intraoperative period and the first 48 hours postoperatively will be abstracted from the medical record.
Changes in Sleep - PSQI | Baseline and 1 month postoperatively
  Changes in sleep will be measured by the Pittsburgh Sleep Quality Index (PSQI) which measures quality and patterns of sleep during the past month. This will be completed at baseline and 1 month postoperatively.
Changes in Sleep - PROMIS | Baseline through 1 month postoperatively
  Changes in sleep will be measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance and Sleep Related Impairment questionnaires. The PROMIS sleep questionnaires assess self-reported perceptions of sleep quality and sleep impairment and will be completed weekly from baseline through 1 month postoperatively.
Biomarkers of inflammation | Baseline, preoperatively, and Day 2 postoperatively
  Blood will be collected at baseline and on postoperative Day 2 to investigate whether the use of a meditation regimen results in a reduction in inflammation and stress secondary to surgery. Subjects randomized to meditation before surgery will also have blood collected preoperatively. Specimens will be frozen for analysis at a later date.

CONTACTS AND LOCATIONS:
Overall Officials: Balachundhar Subramaniam, MD, MPH, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Packiasabapathy S, Susheela AT, Mueller A, Patxot M, Gasangwa DV, O'Gara B, Shaefi S, Marcantonio ER, Yeh GY, Subramaniam B. Guided meditation as an adjunct to enhance postoperative recovery after cardiac surgery: study protocol for a prospective randomized controlled feasibility trial. Trials. 2019 Jan 11;20(1):39. doi: 10.1186/s13063-018-3103-8. PMID 30635064